CLINICAL TRIAL: NCT06970418
Title: Sleep Disorders, Chronotype, and Functional Impairment in the Restrictive ADHD Phenotype
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hande Emine Sabah Barış, Medical Resident, Dr. Behcet Uz Children's Hospital
Other Study IDs: 832
Record Dates: First submitted 2025-05-01; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Sleep Disorders, Circadian Rhythm; Quality of Life; Morningness Eveningness Preference
Keywords: ADHD subtypes, Restrictive ADHD, Sleep disorders, Functionality, Morningness Eveningness Preference
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Disorders, Circadian Rhythm; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Predominantly Inattentive Presentation (ADHD-PI): Patients selected via random sampling from patients either newly admitted to the clinic or already under follow-up for ADHD-PI, with no psychotropic medication use in the last 3 months. All participants were primary or secondary school students. ADHD subtype classification was determined based on Diagnostic and Statistical Manual of Mental Disorders-5 criteria following clinical interviews and scale assessments completed by both parents and teachers. Children with comorbid psychiatric or chronic medical conditions and those using psychostimulants were excluded.
- Restrictive Presentation of ADHD: Patients selected via random sampling from patients either newly admitted to the clinic or already under follow-up for ADHD-R, with no psychotropic medication use in the last 3 months. All participants were primary or secondary school students. ADHD subtype classification was determined based on Diagnostic and Statistical Manual of Mental Disorders-5 criteria following clinical interviews and scale assessments completed by both parents and teachers. Children with comorbid psychiatric or chronic medical conditions and those using psychostimulants were excluded.
- control group: The control group consisted of age- and gender-matched children who presented to the Child and Adolescent Psychiatry clinic, were found to have no psychiatric diagnosis after evaluation, and were considered typically developing. Informed consent and assent forms were obtained from all participants and their legal guardians.

SUMMARY:
This study aims to explore chronotype and sleep disturbances in ADHD subtypes and their relation to functional impairment.

DETAILED DESCRIPTION:
The goal of this observational study is to compare morningness-eveningness and sleep disturbances between children diagnosed with Restrictive ADHD (ADHD-R) and those with Predominantly Inattentive ADHD (ADHD-PI), and to examine how these sleep-related features impact functional impairment.The main question it aims to answer is:Are chronotype differences and sleep disturbances associated with greater functional impairment in children with ADHD-R compared to ADHD-PI and typically developing peers?

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 12 years
* Willingness to participate in the study with provided consent
* Diagnosis of ADHD according to the Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version - Turkish adaptation (K-SADS); no comorbid psychiatric diagnosis (except Oppositional Defiant Disorder)
* Presence of 6 or more inattention symptoms accompanied by 5 or fewer hyperactivity/impulsivity symptoms on the Disruptive Behavior Disorders Rating Scale based on Diagnostic and Statistical Manual of Mental Disorders-IV
* No psychotropic medication use in the past 3 months

Exclusion Criteria:

* Families who do not consent to participate in the study
* Children and adolescents with chronic medical conditions and/or currently taking any medications
* Children and adolescents with intellectual disability (mental retardation)
* Children and adolescents with comorbid psychiatric diagnoses
* Presence of a neurological disorder
* History of head trauma

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 70 children diagnosed with ADHD, aged between 7 and 12 years, were included in the study. This group consisted of 34 children with predominantly inattentive presentation (ADHD-PI) and 36 children with restrictive presentation (ADHD-R), who were either making their first visit to the Child and Adolescent Psychiatry outpatient clinics or were being followed up with a diagnosis of ADHD-PI or ADHD-R, and had not used psychotropic medication in the past three months.
  The control group comprised healthy children with similar age and gender distribution, who were evaluated in the Child and Adolescent Psychiatry clinic but did not receive any psychiatric diagnosis following the assessment.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance Scores | At baseline (upon enrollment)
  Total Score on the Children's Sleep Habits Questionnaire (CSHQ) - Short Form Sleep habits and sleep-related problems will be assessed using the Children's Sleep Habits Questionnaire (CSHQ) - Short Form, a 33-item parent-report measure. Items are rated based on the child's behavior over the past week. Each item is scored from 1 to 3, with higher scores indicating more frequent sleep problems. Items 32 and 33 are scored on a 0-2 scale, and items 1, 2, 3, 10, 11, and 26 are reverse-coded. The total score ranges from 33 to 97. A score of 41 or higher is considered clinically significant, indicating problematic sleep.
  Time Frame: At baseline (upon enrollment) Units of Measure: Total score (range: 33-97) Interpretation: Higher scores indicate more severe sleep problems.

SECONDARY OUTCOMES:
Chronotype classification and total score on the Children's Chronotype Questionnaire (CCQ) | At baseline (upon enrollment)
  Chronotype preference will be assessed using the Children's Chronotype Questionnaire (CCQ), a parent-report tool adapted from the Munich Chronotype Questionnaire and the Children's Morningness-Eveningness Scale. Items 17-26 determine the chronotype score; items 17, 18, 24, and 25 are reverse-coded. Total scores classify children as morning-type (≤23), intermediate-type (24-32), or evening-type (≥33).
  Units of Measure: Chronotype type; total score (range: 10-40); average sleep duration (hours). Higher scores reflect stronger eveningness preference.

OTHER OUTCOMES:
Functional impairment scores on the Weiss Functional Impairment Rating Scale - Parent Form (WFIRS-P) | At baseline (upon enrollment)
  Functional impairment will be assessed using the Weiss Functional Impairment Rating Scale - Parent Form (WFIRS-P), a 50-item Likert-type questionnaire completed by parents. The scale includes six domains: family, school, life skills, self-concept, social activities, and risky behaviors. Each item is rated from 0 ("never") to 3 ("very often"), based on the child's functioning over the past month. Subscale and total scores are calculated by summing item scores and dividing by the number of completed items. Functional impairment in a domain is defined as either scoring 3 on at least one item, 2 on two items, or having a mean score of 1.5 or higher in that domain. overall functional impairment.
  Higher scores indicate greater functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) including age, sex, diagnosis group (ADHD-R or ADHD-PI), and scores from the CSHQ, CCQ, and WFIRS-P will be shared. Data will be available upon reasonable request to academic researchers with an approved proposal and ethics committee approval.